CLINICAL TRIAL: NCT06053021
Title: Antiplatelet Therapy for Acute Ischemic Stroke Patients With Thrombocytopenia
Brief Title: Antiplatelet Therapy for AIS Patients With Thrombocytopenia
Acronym: PERSIST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PERSIST
Record Dates: First submitted 2023-09-11; First posted 2023-09-25 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-09

CONDITIONS: Acute Ischemic Stroke; Thrombocytopenia
MeSH Terms: conditions — Ischemic Stroke; Thrombocytopenia | interventions — Aspirin; Clopidogrel; Cilostazol; Dipyridamole; Platelet Aggregation Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants will be prescribed antiplatelet agents including aspirin, clopidogrel, cilostazol, and dipyridamole.
  Interventions: Drug: aspirin, clopidogrel, cilostazol, and dipyridamole

INTERVENTIONS:
Drug: aspirin, clopidogrel, cilostazol, and dipyridamole — Participants will be prescribed antiplatelet agents including aspirin, clopidogrel, cilostazol, and dipyridamole.
  Other Names: Antiplatelet Agents

SUMMARY:
The goal of this clinical trial is to test the safety and effectiveness of antiplatelet therapy in acute ischemic stroke (AIS) patients with thrombocytopenia. Participants will be prescribed antiplatelet agents and followed up for 3 months.

DETAILED DESCRIPTION:
Antiplatelet therapy is widely used in non-cardiogenic AIS patients for secondary prevention. However, it may also increase the risk of bleeding complications, especially in patients with thrombocytopenia. The goal of this clinical trial is to test the safety and effectiveness of antiplatelet therapy in acute ischemic stroke (AIS) patients with thrombocytopenia. Participants will be prescribed antiplatelet agents and followed up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Acute ischemic stroke or transient ischemic attack with onset < 7 days
* The last blood routine test before enrollment indicates platelet count < 100 x 10^9 and > 30 x 10^9

Exclusion Criteria:

* Chronic renal dysfunction (GFR < 30ml/min) or severe hepatic injury
* Indications for anticoagulation therapy, e.g. atrial fibrillation
* Myocardial infarction within 6 months before enrollment or received percutaneous coronary intervention in the past
* Have or plan to receive CEA or CAS in the following 3 months
* Life expectancy less than 1 year
* Plan to receive invasive surgery in the following 3 months and have high risk of uncontrollable bleeding
* Pregnant or lactating women
* Individuals identified by researchers as unsuitable for participation in the study due to other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
90-day Composite events | 90 days
  Composite events including ischemic stroke, hemorrhagic stroke, myocardial infarction, major extracranial hemorrhage, and vascular death within 90 days after enrollment

SECONDARY OUTCOMES:
90-day ischemic stroke | 90 days
  Ischemic stroke within 90 days after enrollment
90-day hemorrhagic stroke | 90 days
  Hemorrhagic stroke within 90 days after enrollment
90-day myocardial infarction | 90 days
  Myocardial infarction within 90 days after enrollment
90-day major extracranial hemorrhage | 90 days
  Major extracranial hemorrhage within 90 days after enrollment
90-day non-major bleeding | 90 days
  Non-major bleeding within 90 days after enrollment
90-day vascular death | 90 days
  Vascular death within 90 days after enrollment
90-day all-cause death | 90 days
  All-cause death within 90 days after enrollment
Discharge mRS | Through hospitalization, an average of 7 days
  Modified Rankin scale at discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No